CLINICAL TRIAL: NCT06538428
Title: Studying Some Epigenetic Modifications In Glioblastoma Multiforme and Their Impact On Clinical Outcome
Brief Title: Methylation Patterns of the NUPR1, MGMT, NDRG2, and GLI1 Genes and Their Impact on Therapeutic Outcome of GBM Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: ENREC-ASU 2020-8
Record Dates: First submitted 2024-05-12; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-04

CONDITIONS: GBM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — During maximum safe surgical resection, tumor specimens were surgically retrieved using open stereotactic biopsy technique then preserved in neutral buffered formalin and wrapped in paraffin stained with hematoxylin-eosin (HE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GBM group: 58 primary GBM treatment-naïve Egyptian patients DNA methylation profiling for four genes (MGMT, NUPR1,NDRG2,and GLI1 gene) using EpiTect Methyl II (qPCR) system (Qiagen, Germany).
  Interventions: Genetic: DNA methylation profiling
- NND group: DNA methylation profiling for four genes (MGMT, NUPR1,NDRG2,and GLI1 gene) using EpiTect Methyl II (qPCR) system (Qiagen, Germany).
  Interventions: Genetic: DNA methylation profiling

INTERVENTIONS:
Genetic: DNA methylation profiling — measurement of methylation levels of MGMT, NUPR1,NDRG2,and GLI1 gene

SUMMARY:
The study aimed to investigate the role of promoter methylation of MGMT, NUPR1, NDRG2, and GLI1 genes in glioblastoma multiforme (GBM) patients. Tissue samples were collected from GBM patients and individuals with non-neurooncological diseases (NND). The methylation status of the four genes was analyzed, and the clinical characteristics and survival of GBM patients were evaluated.

DETAILED DESCRIPTION:
Objectives. Elucidate the potential role of methylation levels of the MGMT, NUPR1, NDRG2, and GLI1 genes as epigenetic markers for GBM through measuring and comparing the methylation levels of four genes in GBM and NND samples The study researchers started recruiting participants from September 2020 to October 2022, after receiving research ethical approvals from the Medical Ethical Committees at the National Research Center ID#20110 and from the Research Ethics Committee of Faculty of Pharmacy, Ain Shams University, Cairo, Egypt, serial no.[ENREC-ASU 2020-8].

Informed consents were signed by patients or their first-degree relatives. Study participants either patients or controls were informed with the study problem, aim, and objectives. The study was conducted in accordance with the Declaration of Helsinki Guidelines approved in 2013.

A total of 58 primary GBM treatment-naïve Egyptian patients were recruited from the Clinical Oncology Department, Faculty of Medicine, Ain Shams University Hospital, Cairo, Egypt.

Patients' Inclusion Criteria Adult patients (age > 18 years) with a recent diagnosis of GBM and had a performance level of less than or equal to 2 on the Ester Clinical Oncology Group (ECOG) scale .

Therapeutic Approaches, All GBM patients were evaluated clinically, through a full medical history, physical, and neurological examinations. Brain scan was done to enable the patient to receive standardized therapeutic protocol, which includes the greatest secured surgical removal (if attainable), followed by conventional fractionated radiotherapy (aggregate dosage of 60 gray (Gy), provided 2 Gy per fraction for 30 fractions during six weeks) or hypo-fractionated radiotherapy (45 Gy in 15 fractions during three weeks) alongside concurrent TMZ as chemotherapeutic agent in dose of 75 mg/m2 of body surface area daily until the completion of the radiation therapy with periodical follow-up, then re-evaluated clinically and radiologically, given an adjuvant therapy at total of six cycles of TMZ therapy at a dosage of 150 mg/m2 of body surface area from day one to five for a total of 28 days with closely medical surveillance.

Throughout standard medical monitoring, patients underwent evaluation using gadolinium-enhanced magnetic resonance imaging (Gd-MRI) 45 days following radiotherapy and subsequently every three months or whenever medical proof of neurological deterioration emerged.

The demographic characteristics of 58 GBM patients were extracted from the medical records of the hospital. These included demographic attributes such as age in years [22-88], sex (35 male and 23 female), clinicopathological characteristics including ECOG score, date of initial GBM surgery, extent of tumor resection, and previously mentioned therapeutic approach, and survival outcomes including progression-free survival (PFS) and overall survival (OS).

The NND group comprised 20 sex-matched individuals recruited randomly. The age ranged from 4 to 54 years old, with an equal male-to-female ratio of 10 to 10. Those who were not receiving any medications or suffering from any current or past malignancy.

Methods, Sample Proscessing: Before utilizing any oncological therapeutic approaches, brain specimens were surgically retrieved using open stereotactic biopsy technique then preserved in neutral buffered formalin and wrapped in paraffin stained with hematoxylin-eosin (HE). A panel of neuropathologists then assessed all enrolled samples to confirm the diagnosis in accordance with the 2016 CNS Tumors WHO classification.

Optimizing GBM tissue quality for accurate DNA methylation profiling The following inclusion criteria were used to choose the GBM tissue chunks: a histopathological confirmation of GBM tissue with a minimum of 80% viable malignant cells, as well as archived paraffin-embedded tissue sections must be readily available. The subsequent procedures were carried out on all GBM tissues: Full slice of the formalin-fixed, paraffin-embedded (FFPE) block of GBM tissues were cut at a thickness of 4 microns, and subsequently stained with the standard HE stains to evaluate the viability of the donated malignant tissue. Newly cut, up to 10-um-thick FFPE slices were used to prepare samples for PCR analysis.

DNA extraction DNA was isolated from FFPE samples via a QIAamp FFPE kit (Cat. No. 56404 , Valencia, CA), as directed by the supplier. Purity and concentration were determined via a nono-drop spectrophotometer (Quawell, Q-500, Scribner, USA) through determining the intensity of absorption at 260 and 280 nm and verified on a 1% agarose gel. The isolated DNA samples were kept at -20 0C for subsequent analysis to identify methylation levels of MGMT, NUPR1, NDRG2, and GLI1 geneS.

Detection of MGMT, NUPR1, NDRG2, and GLI1 methylation patterns via Methyl II quantitative PCR Methylation patterns of MGMT, NUPR1, NDRG2, and GLI1 have been detected in DNA-retrieved specimens using the EpiTect Methyl II quantitative polymerase chain reaction (qPCR) system (Qiagen, Germany). This is verified by detecting the amount of extracted DNA that remains following fragmentation using methylation specific restriction enzymes. Subsequently, the remaining DNA was quantified by real-time PCR using specific methylation primers for the targeted genes that contain promoter regions of interest.

3.3.1. Methylation-Specific Restriction Enzyme Digestion technique The procedure was conducted in two phases with certain modifications implemented in our laboratory. In Phase I, the EpiTect Methyl II DNA Restriction Kit (cat. no. 335452 ) was utilized for the reactions. Genomic DNA, which had been previously extracted, was aliquoted into two equivalent portions in 2 separate PCR reaction tubes; one tube had no added restriction enzyme and the other tube had methylation-sensitive restriction enzyme that selectively digests unmethylated DNA. The tubes were then subjected to incubation in a thermal cycler (SureCycler 8800, Agilent, Santa Clara, CA, USA) at 37 °C for 6 hours, followed by incubation at 65 °C for 20 minutes.

3.3.2. Quantitative PCR (qPCR) Analysis The quantification of the remaining genomic DNA samples in each tube was performed in Phase II using a Max3005P qPCR system (Stratagene, Agilent Technologies, CA, USA). To initiate this phase, 5 μL aliquot of the remaining DNA from each tube was mixed with the qPCR master mix (RT2 qPCR SYBR Green/ROX Master Mix, Cat. no. 330520 ). The resulting mixture was then dispensed into a PCR plate containing pre-aliquoted MGMT, NUPR1, NDRG2, and GLI1 methylated and unmethylated primers.

Statistical Analysis The Mann-Whitney U test was used to compare the methylation levels of the four genes across the two groups.

The optimal cut-off points for promoter methylation of the four genes were determined after being plotted on (ROC) curves using the mean% of methylation in each patient. The area under the curve (AUC) and test accuracy were calculated.

Survival data (in months) were calculated from the start of each chemotherapy line to the date of death or last follow-up.. Differences in PFS and OS were compared using Kaplan-Meier survival curves, and the log-rank test was used to determine statistical significance.

The Cox proportional hazards model was used for multivariate survival analysis. Cox regression multivariate analysis was performed using a forward stepwise parameter with a significance of 0.05 for entry and 0.1 for removal of factors significantly associated with OS.

The binary logistic regression model was used to analyze the prognostic significance of the methylation of the four genes; MGMT, NUPR1, GLI1, and NUPR1, sex, age, tumor size, and ECOG with respect to clinical outcomes. The goodness-of-fit of the logistic regression models was evaluated using the Hosmer-Lemeshow test.

A significance level of p value less than 0.05 was chosen. Statistical analysis was performed using Statistical package for social studies software (SPSS) version 27.0 (IBM, Armonk, NY) and R Core Team (2023).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years)
* Recent diagnosis of GBM
* Performance status of less than or equal to 2 on the Ester Clinical Oncology Group
* (ECOG) scale,1)
* Pathologically proven GBM

Exclusion Criteria:

* Other types of cancer,
* HBV
* HCV
* Schistosomiasis
* HCC
* HIV
* Alcohol intake
* Thyroid dysfunction
* Inflammatory diseases
* Cerebrovascular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 58 primary GBM treatment-naïve Egyptian patients were recruited from the Clinical Oncology Department, Faculty of Medicine, Ain Shams University Hospital, Cairo, Egypt.
  The NND group comprised 20 sex-matched individuals recruited randomly. The age ranged from 4 to 54 years old, with an equal male-to-female ratio of 10 to 10. Those who were not receiving any medications or suffering from any current or past malignancy.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
GBM prognosis | two years
  Determine the prognostic and predictive significance of the DNA methylation patterns of the examined genes in Egyptian GBM patients. Using the EpiTect Methyl II PCR Kit, The methylation levels of four genes: MGMT, NUPR1, NDRG2, and GLI1 were measured. Then, using Spearman correlation, their levels were correlated with GBM progression and therapeutic response to the chemotherapeutic drug [temozolomide].

SECONDARY OUTCOMES:
Survival analysis | two years
  Obtained correlation between the studied epigenetic events and survival pattern may hopefully in the future direct the clinician to predict the response to standard treatment and provide a guide for proper management of GBM

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hamdy, PhD, Study Director — Professor of Biochemistry, Biochemistry Dept., Faculty of Pharmacy, ASU
Locations (1):
- Ain shams university hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No